CLINICAL TRIAL: NCT00465114
Title: Minimally-invasive Assessment of Cardiac Output in Severe Preeclampsia: Radial Artery Wave Form Analysis Versus Trans-thoracic Echocardiogram
Brief Title: Minimally-invasive Assessment of Cardiac Output in Severe Preeclampsia
Status: Withdrawn | Type: Observational
Why Stopped: Feasibility issues, only 1 patient recruited.
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Other Study IDs: 07-06; 07-0078-E
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Hemodynamic monitoring
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hemodynamic Monitoring

SUMMARY:
Severe preeclampsia often presents with uncontrolled hypertension and therefore requires close monitoring of blood pressure and cardiac performance.

The purpose of the study is to compare two methods of measuring the performance of the heart in pregnant women: one by ultrasound of the heart, the other by assessing the pulse generated in the blood vessel of the wrist. We hope that the method using pulse analysis will be as effective as ultrasound, which is labour intensive and operator dependant.

DETAILED DESCRIPTION:
Severe preeclampsia often presents with uncontrolled hypertension, which requires close monitoring of blood pressure and cardiac output. It will be very useful to know the cardiac output in this patient population, because it will guide the choice of antihypertensive drugs and measure their effect on cardiac output.

Traditionally pulmonary artery catheters were used to measure cardiac output. There are numerous problems with using this method in severe preeclampsia. These include technical difficulty inserting the catheter in an awake, edematous pregnant patient, potentially causing a pneumothorax, damaging the carotid artery or insertion site infection. There is also an increased risk for cardiac arrhythmias. Apart from the risks, the accuracy of the thermodilution measurements can be influenced by factors such as timing of the injection within the respiratory cycle, temperature of the injectate, speed of injection, and placement of the catheter. A readily available, accurate non-invasive cardiac output measurement technique, that will provide reliable data with fewer risks, is needed.

Doppler ultrasound (trans thoracic echocardiography) is the gold standard for measuring cardiac output non-invasively in pregnant patients. Unfortunately the method is operator dependant, not continuous and not always available when needed most.

Recently a device called the FloTrac has been introduced that measures cardiac output minimally invasively. Attached to an arterial line it measures cardiac output every 20 seconds via arterial waveform analysis. The standard of care for measuring blood pressure in severe preeclampsia requires the placement of an intra-arterial line. This group of patients is therefore ideal for measuring cardiac output with the FloTrac, especially since powerful intravenous anti-hypertensives are used to control blood pressure.

Our hypothesis is that the FloTrac will be comparable to Doppler Ultrasound for measuring cardiac output in severely preeclamptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe Preeclampsia
* Arterial Line Required
* Candidates for magnesium sulfate, labetalol or hydrazine

Exclusion Criteria:

* Preexisting cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-04; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada